CLINICAL TRIAL: NCT02600559
Title: An 8-Week, Prospective, Multicenter, Open-Label Study of OTO-201 Given as a Single Administration in Pediatric Subjects With a History of Otitis Media Requiring Tympanostomy Tubes
Brief Title: Open-Label Study of OTO-201 in Pediatric Subjects With a History of Otitis Media Requiring Tympanostomy Tubes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otonomy, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201-201507
Record Dates: First submitted 2015-11-05; First posted 2015-11-09 (Estimated); Results first posted 2020-09-22 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-09

CONDITIONS: Otitis Media
Keywords: Otitis media; Ear infection; Tympanostomy tubes
MeSH Terms: conditions — Otitis Media; Otitis | interventions — Ciprofloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 0.1 mL OTO-201 (Experimental): Ciprofloxacin
  Interventions: Drug: OTO-201 (ciprofloxacin)

INTERVENTIONS:
Drug: OTO-201 (ciprofloxacin)
  Other Names: OTIPRIO

SUMMARY:
This is an 8-week, multicenter, open-label study in which eligible subjects with a history of otitis media requiring TT placement will receive 6 mg OTO-201 to each ear. The study is designed to evaluate the safety and efficacy of OTO-201 in subjects undergoing TT placement with common concurrent surgeries and any middle ear effusion status.

ELIGIBILITY:
Inclusion Criteria includes, but is not limited to:

* Subject is a male or female aged 6 months to 17 years, inclusive
* Subject has a history of otitis media requiring bilateral tympanostomy tube placement
* Subject's caregiver is willing to comply with the protocol and attend all study visits

Exclusion Criteria includes, but is not limited to:

* Subject has a history of prior ear or mastoid surgery, not including myringotomy or myringotomy with TT placement
* Subject has been designated for any other surgical procedure that would occur concurrently with TT placement, except adenoidectomy, airway endoscopy, nasal endoscopy, and nasal cautery for epistaxis
* Subject has a history of sensorineural hearing loss

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 501 (Actual)
Dates: Start 2015-10; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dean Hakanson, MD, Study Chair — Otonomy, Inc.
Locations (1):
- Email Otonomy Central Contact for Trial Locations, San Diego, California, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were a total of 518 subjects screened for this study. There were 17 subjects considered screen failures, with the majority (11) failing to meet inclusion/exclusion criteria. Therefore, 501 subjects were assigned for treatment in this study and are designated as "enrolled".
Groups:
- 6 mg OTO-201: 6 mg ciprofloxacin: single administration
Period: Overall Study
Arm/Group | 6 mg OTO-201
Started | 501
Completed | 478
Not Completed | 23
Not completed — Withdrawal by Subject | 3
Not completed — Lost to Follow-up | 20

BASELINE CHARACTERISTICS:
Arm/Group | 6 mg OTO-201
Number analyzed (Participants) | 501
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 501
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 2.9 (2.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 216
  Male | 285
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 80
  Not Hispanic or Latino | 403
  Unknown or Not Reported | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 6
  Native Hawaiian or Other Pacific Islander | 3
  Black or African American | 40
  White | 415
  More than one race | 0
  Unknown or Not Reported | 36
Region of Enrollment [Number; unit: participants]
  United States | 501
Medicaid (Yes/No) [Count of Participants; unit: Participants]
  Medicaid - Yes | 165
  Medicaid - No | 336

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Post-surgical Otorrhea
Description: Absence or presence of otorrhea (drainage from the middle ear)
Time Frame: Week 4
Population: Safety analysis set: All subjects who received study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | 6 mg OTO-201
Number analyzed (Participants) | 501
Participants
  Absence of Otorrhea | 383
  Presence of Otorrhea | 118

2. Primary Outcome: Number of Subjects With Post-surgical Otorrhea
Description: Absence or presence of otorrhea (drainage from the middle ear)
Time Frame: 8 weeks
Population: Safety analysis set: All subjects who received study drug
Measure: Count of Participants; unit: Participants
Arm/Group | 6 mg OTO-201
Number analyzed (Participants) | 501
Participants
  Absence of Otorrhea | 334
  Presence of Otorrhea | 167

3. Secondary Outcome: Adverse Events
Description: Evaluation of adverse events
Time Frame: Up to Eight Weeks
Population: Safety analysis set: All subjects who received study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | 6 mg OTO-201
Number analyzed (Participants) | 501
Participants
  Subjects with AEs | 250
  Subjects without AEs | 251

4. Secondary Outcome: Caregiver Burden - Ear Discharge Control
Description: Ear Drop Caregiver Burden Questionnaire at Week 4
Time Frame: Week 4
Population: Safety analysis set: All subjects who received study drug and whose caregiver completed the questionnaire at Week 4
Measure: Count of Participants; unit: Participants
Arm/Group | 6 mg OTO-201
Number analyzed (Participants) | 485
Participants
  Satisfied with control of ear discharge | 481
  Not satisfied with control of ear discharge | 4

5. Secondary Outcome: Caregiver Burden - Ear Discharge Control
Description: Ear Drop Caregiver Burden Questionnaire at Week 8
Time Frame: Week 8
Population: Safety analysis set: All subjects who received study drug, and had a completed questionnaire at Week 8
Measure: Count of Participants; unit: Participants
Arm/Group | 6 mg OTO-201
Number analyzed (Participants) | 475
Participants
  Satisfied with control of ear discharge | 470
  Not satisfied with control of ear discharge | 5

6. Secondary Outcome: Caregiver Burden - Ear Drops Administration
Description: Ear Drop Caregiver Burden Questionnaire at Week 8
Time Frame: Week 8
Population: Safety analysis set: All subject who received study drug, and who had to be treated with ear drops after tube placement surgery.
Measure: Count of Participants; unit: Participants
Arm/Group | 6 mg OTO-201
Number analyzed (Participants) | 71
Participants
  Bothersome to administer ear drops | 48
  Not bothersome to administer ear drops | 23

ADVERSE EVENTS:
Time Frame: Adverse events were reported during dosing and up to 2 months following tympanostomy tube surgery.
Arm/Group | 6 mg OTO-201
All-Cause Mortality (participants affected / at risk) | 0/501
Serious Adverse Events (participants affected / at risk) | 1/501
Other Adverse Events (participants affected / at risk) | 200/501
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 6 mg OTO-201 (N=501)
Influenza (Infections and infestations) | 1 (501) — One of 4 adverse events that caused the subject to be hospitalized (also pneumonia, rhinovirus infection, and streptococcal infection); not related to study drug.
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 6 mg OTO-201 (N=501)
Upper Respiratory Infection (Infections and infestations) | 35
Nasopharyngitis (Infections and infestations) | 13
Sinusitis (Infections and infestations) | 12
Otitis Media (Infections and infestations) | 11
Pharyngitis streptococcal (Infections and infestations) | 8
Device occlusion (General disorders) | 67
Pyrexia (General disorders) | 41
Device extrusion (General disorders) | 9
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 19
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 12
Ear Pain (Ear and labyrinth disorders) | 26
Vomiting (Gastrointestinal disorders) | 12
Procedural pain (Injury, poisoning and procedural complications) | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication subject to Sponsor consent.